CLINICAL TRIAL: NCT02854228
Title: PITUItary Carcinomas or Aggressive Tumors REgistry: Monocentric Study Form a Cohort of Patient Operated on for Pituitary Tumors in University Hospital of Lyon (France)
Brief Title: PITUItary Carcinoma or Aggressive Tumors REgistry -Lyon
Acronym: PITUICARE-Lyon
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0506
Record Dates: First submitted 2016-07-27; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Pituitary Tumor
Keywords: Pituitary tumor; pituitary carcinoma; acromegaly; cushing; prolactinoma
MeSH Terms: conditions — Pituitary Neoplasms; Acromegaly; Prolactinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA and pituitary tumor frozen sample (Neurobiotec Biological Resource Centre (BRC) of Hospices Civils de Lyon (HCL))
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to observe predictors of pituitary tumor recurrence and markers of persistent disease activity through computerized collection of comprehensive demographic, therapeutic, pathologic and outcome information on patients harboring pituitary mass lesions of all types.

ELIGIBILITY:
Inclusion Criteria:

• patients with confirmed pituitary disease

Exclusion Criteria:

• patients who do not have confirmed pituitary disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: tertiary referral center
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2007-02; Primary Completion 2015-12 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival after pituitary surgery according to the clinicopathological classification (HYPOPRONOS) | up to 10 years (postoperatively)
  Clinical, biochemical et imaging evaluation of a cohort of patient operated in the referral center for pituitary tumor.
  Identification of recurrence or progression an analysis of the clinicopathological classification.
  Evaluation of the different therapeutic strategies (med, surgery, chemotherapies, radiation therapy) to prevent recurrence or tumor progression.

SECONDARY OUTCOMES:
Correlation between percentage of SSTR expression of the pituitary tumor and somatostatine analogs efficacy. | 2007-2020
  Analysis of the expression of SST receptors in GH, PRL and ACTH secreting pituitary tumors: SSTR expression accessed by immunohistochemistry of the pituitary tumor.
  Evaluation of the response to somatostatine analogs: somatostatine analogs efficacy evaluated by normalization of hormone hypersecretion in ACTH, GH and PRL secreting pituitary tumor.
Correlation between percentage of MGMT expression of the pituitary tumor and tumor response to temozolomide. | 2007-2020
  Evaluation of MGMT expression (accessed by immunohistochemistry of the pituitary tumor) and response to temozolomide treatment (evaluated according to RECIST criteria) for patient presenting multirecurrent tumors resistant to conventional treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Raverot, MD PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Groupement Hospitalier Est, Lyon, France, Bron, France

REFERENCES:
- [Derived] Raverot G, Dantony E, Beauvy J, Vasiljevic A, Mikolasek S, Borson-Chazot F, Jouanneau E, Roy P, Trouillas J. Risk of Recurrence in Pituitary Neuroendocrine Tumors: A Prospective Study Using a Five-Tiered Classification. J Clin Endocrinol Metab. 2017 Sep 1;102(9):3368-3374. doi: 10.1210/jc.2017-00773. PMID 28651368